CLINICAL TRIAL: NCT02445001
Title: Erythrocyte Ghost Mediated Retinal Diagnosis
Acronym: EGMRetinalDx
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn before recruitment started.
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-163A
Record Dates: First submitted 2013-10-28; First posted 2015-05-15 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICG loaded erythrocytes (Experimental): Ability to directly visualize erythrocyte dynamics within the retinal and choroidal microcirculations would facilitate focused investigations into the relationships between vasomotion (i.e., pulsatile erythrocyte movement through capillaries) and oxygen distribution to localized tissue regions.
  Interventions: Procedure: ICG loaded erythrocytes

INTERVENTIONS:
Procedure: ICG loaded erythrocytes — For each subject, on the morning of the day angiography was scheduled, or no longer than 4 days prior to angiography, 9 ml of blood will be withdrawn from an antecubital vein. Using sterile procedures, erythrocyte ghosts produced from the blood will be loaded with ICG dye (for the diagnostic part of the study) or with ICG and one of several drugs (for the therapeutic part of the study) by the following procedure, which requires about 2 hours and yields approximately 1 ml of packed cells (80% Ht) that, after microscopic examination, are ready for autologous re-injection
  Other Names: Erythrocyte mediated diagnostic angiography

SUMMARY:
Instead of the usual procedure of injecting ICG dye directly into an arm vein, now the dye can be placed inside of RBCs. When a small volume of the RBC's with the dye is injected into a person's arm, the individual RBCs can be seen as they flow through the retinal blood vessels.

DETAILED DESCRIPTION:
Capillary erythrocyte movement throughout the entire human macula can be observed routinely for periods up to 20 minutes by autologous re-injection of a small volume (about 1 mL) of indocyanine green (ICG)-loaded erythrocytes, making possible for the first time quantification of blood flow in individual capillaries, including abnormal structures like choroidal neovascularization (CNV), and it makes possible characterization of vasomotion in ocular vasculatures.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female, of any race who is at least 40 years of age and has clinical signs of CNV or exudative manifestations of AMD, has clinical signs of DR, or clinical signs of retinal occlusive disease.
2. Patients with subfoveal, extrafoveal or juxtafoveal CNV, which is classic, minimally classic or occult and has dimensions less than 25.0 mm2 as measured on the sodium fluorescein angiogram (SFA).
3. Patient with recurrent CNV, where previous treatment never involved the foveal avascular zone (FAZ).
4. Analysis of highspeed ICGA must show one or more welldefined feeder vessel.
5. Patient must have best corrected visual acuity based on the ETDRS chart between 20/40 and 20/320 in the study eye.
6. Patient must be willing, be able to comply with the protocol and provide informed consent.

Exclusion Criteria:

1. CNV secondary to any cause other than AMD or DR.
2. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
3. Patient participating in any other investigational drug study.
4. Patient with significant liver disease or uremia.
5. Patient with known adverse reaction to indocyanine green or iodine.
6. Patient is pregnant or nursing.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Capillary erythrocyte movement | 1 hour
  To demonstrate in each subject eye the differences between erythrocyte movement through retinal and choroidal capillaries in normal fundus areas and their movement through abnormal areas associated with vascular disease

SECONDARY OUTCOMES:
Retinal capillary movement | 1 hour
  To demonstrate the relationship between the state of retinal vasomotion and retinal edema in the human eye. The primary focus will be on eyes with CNV associated with age-related macular degeneration (AMD) and eyes with diabetic retinopathy (DR).

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Yannuzzi, MD, Principal Investigator — NSLIJ/MEETH
Locations (1):
- Northshore LIJ/MEETH Campus, New York, New York, United States

REFERENCES:
- [Background] Flower RW. Experimental studies of indocyanine green dye-enhanced photocoagulation of choroidal neovascularization feeder vessels. Am J Ophthalmol. 2000 Apr;129(4):501-12. doi: 10.1016/s0002-9394(99)00411-0. PMID 10764860